CLINICAL TRIAL: NCT02266732
Title: Ultrasound Vs Nerve Stimulation - Why is a PNS so Effective?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN11/9771; 11/YH/0206 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-10-03; First posted 2014-10-17 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

ARMS (2):
- Interscalene block (Other)
  Interventions: Device: Stimuplex HNS 12
- Femoral block (Other)
  Interventions: Device: Stimuplex HNS 12

INTERVENTIONS:
Device: Stimuplex HNS 12
  Other Names: Peripheral nerve stimulator for nerve location

SUMMARY:
The traditional model of localizing a nerve for blockade is using a peripheral nerve stimulator, PNS. Recent advances in UltraSound technology has allowed UltraSound to guide nerve blockade. However despite excellent visualization nerve block success has not significantly improved. I aim to show that this is because the PNS stimulation of a nerve is more than a proximity response as thought but a correct fascial plane response and hence the high success rate of this blind approach.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 to 3 patients for any shoulder surgery or unilateral ACL knee surgery

Exclusion Criteria:

* Refusal to consent
* Allergy to Chirocaine local anaesthetic
* Pace maker in situ
* Sepsis at site of regional block

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Nerve stimulation resulting in muscle contraction or not | Five minutes
  Whether the nerve is successfully stimulated, resulting in muscle contraction, or not when the needle is on the wrong side of the fascial layer.